CLINICAL TRIAL: NCT00350532
Title: Clonidine-induced Spinal Acetylcholine Release: Normal Volunteers vs. Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01NS041386_TRIAL2; P01NS041386 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: pain, chronic pain; acetylcholine; clonidine; a2-adrenergic agonists; alpha2-adrenergic agonists
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neuropathic Pain Subjects (Active Comparator): Chronic Pain Participants will be trained to accurately estimate pain by way of thermal heat testing. Next a small amount of spinal fluid will be withdrawn from each participant to measure the amounts of naturally-made chemicals in the participants' cerebrospinal fluid. Participants then will receive an injection of clonidine. After the injection, additional samples of spinal fluid will be taken to measure chemical changes in the fluid.
  Interventions: Drug: clonidine
- Healthy Subjects (Active Comparator): Healthy Participants will be trained to accurately estimate pain by way of thermal heat testing. Next a small amount of spinal fluid will be withdrawn from each participant to measure the amounts of naturally-made chemicals in the participants' cerebrospinal fluid. Participants then will receive an injection of clonidine. After the injection, additional samples of spinal fluid will be taken to measure chemical changes in the fluid.
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — Patients will receive intrathecal clonidine (or clonidine injected into cerebrospinal fluid)
  Arms: Neuropathic Pain Subjects
Drug: clonidine — Patients will receive intrathecal clonidine (or clonidine injected into cerebrospinal fluid)
  Arms: Healthy Subjects

SUMMARY:
The purpose of this study is to compare the amount of acetylcholine release after a single injection of clonidine in normal volunteers and individuals with neuropathic pain.

DETAILED DESCRIPTION:
This study is part of a pain center grant that focuses on how pain, especially chronic neuropathic pain, alters the response to traditional and non-traditional analgesics (pain medications).

The way that nerve fibers carry pain information to the brain is thought to change after surgery and in cases of chronic pain. For this reason, some medicines work better to relieve pain in healthy people who have a sudden painful injury when compared to people after surgery or to people with chronic pain. Currently available pain medications may not relieve all types of pain or may relieve pain only at doses that produce side effects and potential complications.

The aim of this study is to understand the mechanisms by which intrathecal clonidine (or clonidine injected into cerebrospinal fluid) increases in potency and efficacy by examining the cerebrospinal fluid of healthy individuals, before and after clonidine administration, as well as looking at the spinal fluid of people with chronic neuropathic nerve pain. More specifically, in this study, researchers will compare acetylcholine release (a protein-like substance found in cerebrospinal fluid) in normal volunteers and patients with neuropathic pain after a single injection of clonidine.

After baseline measurements, including blood pressure and heart rate, participants will be trained to accurately estimate pain by way of thermal heat testing. Next a small amount of spinal fluid will be withdrawn from each participant to measure the amounts of naturally-made chemicals in the participants' cerebrospinal fluid. Participants then will receive an injection of clonidine. After the injection, additional samples of spinal fluid will be taken to measure chemical changes in the fluid.

Duration of the study for participants is 1 day, and includes 1 visit to the research center, lasting approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* Patients with neuropathic pain

Exclusion Criteria:

* Pregnancy
* Allergy to clonidine
* Currently taking clonidine or other direct a2-adrenergic agonists
* Taking cholinesterase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences; Richard Rauck, M.D., Principal Investigator — The Center for Clinical Research
Locations (2):
- United States (2):
  - The Center for Clinical Research, 145 Kimel Park Drive, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Medical Center Boulevard, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9/1/2004-6/2/2006. Subjects were recruited from a pain clinic and the control group were healthy subjects.
Pre-assignment Details: No significant events or abnormal approaches noted.
Groups:
- Neuropathic Pain Subjects; Healthy Subjects: Participants will be trained to accurately estimate pain by way of thermal heat testing. Next a small amount of spinal fluid will be withdrawn from each participant to measure the amounts of naturally-made chemicals in the participants' cerebrospinal fluid. Participants then will receive an injection of clonidine. After the injection, additional samples of spinal fluid will be taken to measure chemical changes in the fluid.
Period: Overall Study
Arm/Group | Neuropathic Pain Subjects | Healthy Subjects
Started | 24 | 19
Completed | 24 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Neuropathic Pain Subjects: Subjects with existing neuropathic pain Outcome criterion is acetylcholine concentration in cerebrospinal fluid (CSF) at 60 minutes after injection.
- Healthy Subjects: Healthy subjects with no existing pain conditions. Outcome criterion is acetylcholine concentration in cerebrospinal fluid (CSF) at 60 minutes after injection.
- Total: Total of all reporting groups
Arm/Group | Neuropathic Pain Subjects | Healthy Subjects | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 19 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.875 (11.48) | 32 (8.51) | 40.86 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Acetylcholine Concentration in Cerebrospinal Fluid
Description: Acetylcholine levels in CSF after administration of intrathecal clonidine measured by High-performance liquid chromatography (HPLC).
Time Frame: 60 minutes
Population: There was no difference noted in acetylcholine levels in healthy subjects compared to subjects with chronic pain
Measure: Mean (Full Range); unit: picograms per milliliter (pg/ml)
Arm/Group | Neuropathic Pain Subjects | Healthy Subjects
Number analyzed (Participants) | 24 | 19
picograms per milliliter (pg/ml) | 406 [383 to 406] | 383 [383 to 406]

ADVERSE EVENTS:
Arm/Group | Neuropathic Pain Subjects | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/19
Other Adverse Events (participants affected / at risk) | 0/24 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No